CLINICAL TRIAL: NCT00818324
Title: Long Term Administration Study of OPC-12759 Ophthalmic Suspension in Dry Eye Patients
Brief Title: Long Term Administration Study of OPC-12759 Ophthalmic Suspension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Eiji Murakami/Director of Division of Dermatologicals and Ophthalmologicals, Otsuka Pharmaceutical Co., Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 037E-08-002
Record Dates: First submitted 2009-01-04; First posted 2009-01-07 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-01

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-12759 Ophthalmic suspension (Experimental): Instillation, 4times/day
  Interventions: Drug: OPC-12759 Ophthalmic suspension

INTERVENTIONS:
Drug: OPC-12759 Ophthalmic suspension — Instillation,4times/day,for 52weeks

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of OPC-12759 ophthalmic suspension during 52 weeks in dry eye patients

ELIGIBILITY:
Inclusion Criteria:

1. Out patient;
2. Ocular discomfort severity is moderate to severe;
3. Corneal-conjunctival damage is moderate to severe;
4. Unanesthetized Schirmer's test score of 5mm/5minutes or less,or tear breakup time is 5 seconds or less;
5. Best corrected visual acuity of 0.2 or better in both eyes.

Exclusion Criteria:

1. Presence of anterior segment disease or disorder other than that associated with keratoconjunctivitis scicca;
2. Ocular hypertention patient or glaucoma patient with ophthalmic solution;
3. Anticipated use of any topically-instilled ocular medications or patients who cannot discontinue the use during the study;
4. Anticipated use of contact lens during the study;
5. Patient with punctal plug;
6. Any history of ocular surgery within 12 months;
7. Female patients who are pregnant, possibly pregnant or breast feeding;
8. Known hypersensitivity to any component of the study drug or procedual medications;
9. Receipt of any investigational product within 4 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Murakami, Study Chair — OPCJ-DDO
Locations (5):
- Japan (5):
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Tohoku Region
  - Tokai Region

RESULTS

PARTICIPANT FLOW:
Groups:
- 2% Rebamipide Group: 2% rebamipide ophthalmic suspension received one drop of to both eyes four times a day for 52 weeks
Period: Overall Study
Arm/Group | 2% Rebamipide Group
Started | 154
Completed | 127
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | 2% Rebamipide Group
Number analyzed (Participants) | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (14.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 15
Region of Enrollment [Number; unit: participants]
  Japan | 154

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFB) in Fluorescein Corneal Staining (FCS) Score
Description: FCS indicates the damage to the corneal epithelium. Per the National Eye Institute/Industry Workshop report, the cornea was divided into 5 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated (0-15). 0 is better. Baseline scores and those obtained at each examination time point were compared (paired t-test).
Time Frame: Baseline, Week2, Week4, Week28, Week52
Measure: Mean (Standard Deviation); unit: FCS score
Arm/Group | 2% Rebamipide Group
Number analyzed (Participants) | 154
FCS score
  CFB at Week2 (n=154) | -2.2 (2.3)
  CFB at Week4 (n=149) | -2.7 (2.4)
  CFB at Week28 (n=135) | -4.1 (2.8)
  CFB at Week52 (n=127) | -4.6 (2.6)
Statistical Analysis 1: Comparison: 2% Rebamipide Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The p value represents the comparison between baseline data and data at Week 2
Statistical Analysis 2: Comparison: 2% Rebamipide Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The p value represents the comparison between baseline data and data at Week 4
Statistical Analysis 3: Comparison: 2% Rebamipide Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The p value represents the comparison between baseline data and data at Week 28
Statistical Analysis 4: Comparison: 2% Rebamipide Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The p value represents the comparison between baseline data and data at Week 52

2. Other Pre Specified Outcome: Change From Baseline (CFB) in Lissamine Green Conjunctival Staining (LGCS) Score
Description: LGCS indicates the damage to the conjunctival epithelium. Per the National Eye Institute/Industry Workshop report, the conjunctiva was divided into 6 fractions, each of which was given a staining score from 0 to 3, and the total score was calculated (0-18). 0 is better. Baseline scores and those obtained at each examination time point were compared (paired t-test).
Time Frame: Baseline, Week2, Week4, Week28, Week52
Measure: Mean (Standard Deviation); unit: LGCS score
Arm/Group | 2% Rebamipide Group
Number analyzed (Participants) | 154
LGCS score
  CFB at Week2 (n=154) | -2.6 (3.0)
  CFB at Week4 (n=149) | -3.3 (3.2)
  CFB at Week28 (n=135) | -5.7 (4.0)
  CFB at Week52 (n=127) | -6.0 (3.7)
Statistical Analysis 1: Comparison: 2% Rebamipide Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The p value represents the comparison between baseline data and data at Week 2
Statistical Analysis 2: Comparison: 2% Rebamipide Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The p value represents the comparison between baseline data and data at Week 4
Statistical Analysis 3: Comparison: 2% Rebamipide Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The p value represents the comparison between baseline data and data at Week 28
Statistical Analysis 4: Comparison: 2% Rebamipide Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The p value represents the comparison between baseline data and data at Week 52

ADVERSE EVENTS:
Time Frame: 52 Weeks
Arm/Group | 2% Rebamipide Group
Serious Adverse Events (participants affected / at risk) | 6/154
Other Adverse Events (participants affected / at risk) | 125/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2% Rebamipide Group (N=154)
Hypothyroidism (Endocrine disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Surgical vascular shunt (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2% Rebamipide Group (N=154)
Abnormal sensation in eye (Eye disorders) | 3 (3)
Blepharitis (Eye disorders) | 5 (5)
Conjunctival haemorrhage (Eye disorders) | 8 (8)
Conjunctivitis (Eye disorders) | 7 (7)
Conjunctivitis allergic (Eye disorders) | 8 (8)
Dry eye (Eye disorders) | 2 (2)
Eye discharge (Eye disorders) | 5 (5)
Eye irritation (Eye disorders) | 6 (6)
Eye pain (Eye disorders) | 4 (4)
Lacrimation decreased (Eye disorders) | 2 (2)
Lacrimation increased (Eye disorders) | 2 (2)
Retinal haemorrhage (Eye disorders) | 3 (3)
Trichiasis (Eye disorders) | 8 (8)
Vision blurred (Eye disorders) | 5 (5)
Visual acuity reduced (Eye disorders) | 4 (4)
Foreign body sensation in eyes (Eye disorders) | 2 (2)
Conjunctival hyperaemia (Eye disorders) | 5 (5)
Meibomian gland discharge (Eye disorders) | 2 (2)
Eye pruritus (Eye disorders) | 2 (2)
Ocular discomfort (Eye disorders) | 3 (3)
Dacryostenosis acquired (Eye disorders) | 2 (2)
Corneal disorder (Eye disorders) | 4 (4)
Meibomian gland dysfunction (Eye disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5)
Dental caries (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Periodontitis (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Cystitis (Infections and infestations) | 4 (4)
Dacryocystitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 34 (34)
Urinary tract infection (Infections and infestations) | 2 (2)
Conjunctivitis bacterial (Infections and infestations) | 3 (3)
Foreign body in eye (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 6 (6)
Blood urea increased (Investigations) | 5 (5)
Gamma-glutamyltransferase increased (Investigations) | 3 (3)
Glucose urine present (Investigations) | 4 (4)
White blood cell count decreased (Investigations) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (bitter taste) (Nervous system disorders) | 21 (21)
Headache (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Peripheral coldness (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No